CLINICAL TRIAL: NCT05499520
Title: Project RESIST: Evaluating the Effects of Anti-smoking Inoculation Messages Among Young Adult Sexual Minority Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Harvard School of Public Health (HSPH) (Other); Stanford University (Other); Dana-Farber Cancer Institute (Other); Fenway Community Health (Other)
Responsible Party: Principal Investigator, Andy Tan, Associate Professor, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 11022; R01CA237670 (NIH)
Record Dates: First submitted 2022-08-04; First posted 2022-08-12 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cigarette Smoking Behavior
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- Currently Smoking, No Message Condition (No Intervention): Participants will receive no anti-smoking messages. They will receive the threat message during the baseline survey. Outcomes will be measured before and immediately after seeing the threat message, and at 1 month.
- Currently Smoking, Single Message Immediate (Experimental): Participants will receive a single anti-smoking message followed by the threat message during the baseline survey. Outcomes will be measured before seeing the anti-smoking message and threat message, immediately after seeing the threat message, and at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages
- Currently Smoking, Single Message 1 Week Delay (Experimental): Participants will receive a single anti-smoking message during the baseline survey, followed by the threat message one week later in a separate survey. Outcomes will be measured before seeing the anti-smoking message at baseline, immediately after seeing the threat message at 1 week, and at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages
- Currently Smoking, Single Message 1 Month Delay (Experimental): Participants will receive a single anti-smoking message during the baseline survey, followed by the threat message one month later in a separate survey. Outcomes will be measured before seeing the anti-smoking message at baseline, and immediately after seeing the threat message at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages
- Currently Smoking, Single Message 1 Month Delay, Repeated Exposure (Experimental): Participants will receive a single anti-smoking message during the baseline survey, followed by the threat message one month later. Participants will also receive repeated exposures of a single anti-smoking message at 1, 2, and 3 weeks in separate surveys. Outcomes will be measured before seeing the anti-smoking message at baseline and immediately after seeing the threat message at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages
- Currently Smoking, Three Messages Immediate (Experimental): Participants will receive three anti-smoking messages, followed by the threat message during the baseline survey. Outcomes will be measured before seeing the anti-smoking messages and threat message, immediately after seeing the threat message, and at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages
- Currently Smoking, Three Messages 1 Week Delay (Experimental): Participants will receive three anti-smoking messages during the baseline survey, followed by the threat message one week later in a separate survey. Outcomes will be measured before seeing the anti-smoking messages at baseline, immediately after seeing the threat message at 1 week, and at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages
- Currently Smoking, Three Messages 1 Month Delay (Experimental): Participants will receive three anti-smoking messages during the baseline survey, followed by the threat message one month later in a separate survey. Outcomes will be measured before seeing the anti-smoking messages at baseline, and immediately after seeing the threat message at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages
- Currently Smoking, Three Messages 1 Month Delay Repeat Exposure (Experimental): Participants will receive three anti-smoking messages during the baseline survey, followed by the threat message one month later. Participants will also receive repeated exposures of three anti-smoking messages at 1, 2, and 3 weeks in separate surveys. Outcomes will be measured before seeing the anti-smoking messages at baseline and immediately after seeing the threat message at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages
- Not Currently Smoking, No Message Condition (No Intervention): Participants will receive no anti-smoking messages. They will receive the threat message during the baseline survey. Outcomes will be measured before and immediately after seeing the threat message, and at 1 month.
- Not Currently Smoking, Single Message Immediate (Experimental): Participants will receive a single anti-smoking message followed by the threat message during the baseline survey. Outcomes will be measured before seeing the anti-smoking message and threat message, immediately after seeing the threat message, and at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages
- Not Currently Smoking, Single Message 1 Week Delay (Experimental): Participants will receive a single anti-smoking message during the baseline survey, followed by the threat message one week later in a separate survey. Outcomes will be measured before seeing the anti-smoking message at baseline, immediately after seeing the threat message at 1 week, and at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages
- Not Currently Smoking, Single Message 1 Month Delay (Experimental): Participants will receive a single anti-smoking message during the baseline survey, followed by the threat message one month later in a separate survey. Outcomes will be measured before seeing the anti-smoking message at baseline, and immediately after seeing the threat message at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages
- Not Currently Smoking, Single Message 1 Month Delay, Repeated Exposure (Experimental): Participants will receive a single anti-smoking message during the baseline survey, followed by the threat message one month later. Participants will also receive repeated exposures of a single anti-smoking message at 1, 2, and 3 weeks in separate surveys. Outcomes will be measured before seeing the anti-smoking message at baseline and immediately after seeing the threat message at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages
- Not Currently Smoking, Three Messages Immediate (Experimental): Participants will receive three anti-smoking messages, followed by the threat message during the baseline survey. Outcomes will be measured before seeing the anti-smoking messages and threat message, immediately after seeing the threat message, and at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages
- Not Currently Smoking, Three Messages 1 Week Delay (Experimental): Participants will receive three anti-smoking messages during the baseline survey, followed by the threat message one week later in a separate survey. Outcomes will be measured before seeing the anti-smoking messages at baseline, immediately after seeing the threat message at 1 week, and at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages
- Not Currently Smoking, Three Messages 1 Month Delay (Experimental): Participants will receive three anti-smoking messages during the baseline survey, followed by the threat message one month later in a separate survey. Outcomes will be measured before seeing the anti-smoking messages at baseline, and immediately after seeing the threat message at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages
- Not Currently Smoking, Three Messages 1 Month Delay Repeat Exposure (Experimental): Participants will receive three anti-smoking messages during the baseline survey, followed by the threat message one month later. Participants will also receive repeated exposures of three anti-smoking messages at 1, 2, and 3 weeks in separate surveys. Outcomes will be measured before seeing the anti-smoking messages at baseline and immediately after seeing the threat message at 1 month.
  Interventions: Other: Culturally Tailored Anti-Smoking Messages

INTERVENTIONS:
Other: Culturally Tailored Anti-Smoking Messages — Anti-smoking messages will be administered online via a Qualtrics survey.
  Arms: Currently Smoking, Single Message 1 Month Delay; Currently Smoking, Single Message 1 Month Delay, Repeated Exposure; Currently Smoking, Single Message 1 Week Delay; Currently Smoking, Single Message Immediate; Currently Smoking, Three Messages 1 Month Delay; Currently Smoking, Three Messages 1 Month Delay Repeat Exposure; Currently Smoking, Three Messages 1 Week Delay; Currently Smoking, Three Messages Immediate; Not Currently Smoking, Single Message 1 Month Delay; Not Currently Smoking, Single Message 1 Month Delay, Repeated Exposure; Not Currently Smoking, Single Message 1 Week Delay; Not Currently Smoking, Single Message Immediate; Not Currently Smoking, Three Messages 1 Month Delay; Not Currently Smoking, Three Messages 1 Month Delay Repeat Exposure; Not Currently Smoking, Three Messages 1 Week Delay; Not Currently Smoking, Three Messages Immediate

SUMMARY:
Project RESIST is an R01 study funded by NCI focused on determining the effects of using culturally tailored inoculation approaches to increase resilience to tobacco marketing influences among young adult sexual minority women ages 18-30 and incorporates critical stakeholder inputs that support later adoption and implementation. The study team is utilizing formative research to design and pre-test anti-smoking messages and two national longitudinal online survey experiments.

DETAILED DESCRIPTION:
This study will recruit 3000 young adult sexual minority women (SMW), ages 18-30 years, current smokers (n = 1500) and not current smokers (n = 1500). The study will determine the effects of varying the dose (single vs. multiple), and latency (immediate vs. delayed) of showing participants inoculation anti-smoking messages on smoking and quitting intentions. The study team hypothesize that the multiple exposures (vs. single), and delayed exposure (vs. immediate) will be associated with increased resistance to marketing, reduced smoking intention, and increased quitting intention. The study team will further explore the mechanisms of inoculation effects through emotions, beliefs, and attitudes towards tobacco companies. Participants will be asked to complete a baseline survey and then will receive an anti-smoking message in varying dosages based on the condition they are assigned with a control group receiving no message. Participants will then see a pro-smoking or threat message immediately, one week, or one month late, depending on the condition they were assigned.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-30
* Woman
* Identifies as a sexual minority (any sexual orientation other than heterosexual)
* Lives in the United States
* Able to take surveys in English

Exclusion Criteria:

* Under 18 or older than 30
* Men
* Heterosexual
* Lives outside the United States
* Unable to take the survey in English

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Anyone who identifies as a woman, whether they are cisgender or transgender, would meet the gender-based eligibility requirement
Enrollment: 2591 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Currently Smoking, No Message Condition; Not Currently Smoking, No Message Condition: Participants will receive no anti-smoking messages. They will receive the threat message during the baseline survey. Outcomes will be measured before and immediately after seeing the threat message.
- Currently Smoking, Single Message Immediate; Not Currently Smoking, Single Message Immediate: Participants will receive a single anti-smoking message followed by the threat message during the baseline survey. Outcomes will be measured before seeing the anti-smoking message and threat message, immediately after seeing the threat message.
  Culturally Tailored Anti-Smoking Messages: Anti-smoking messages will be administered online via a Qualtrics survey.
- Currently Smoking, Single Message 1 Week Delay; Not Currently Smoking, Single Message 1 Week Delay: Participants will receive a single anti-smoking message during the baseline survey, followed by the threat message one week later in a separate survey. Outcomes will be measured before seeing the anti-smoking message at baseline, immediately after seeing the threat message at 1 week.
  Culturally Tailored Anti-Smoking Messages: Anti-smoking messages will be administered online via a Qualtrics survey.
- Currently Smoking, Single Message 1 Month Delay: Participants will receive a single anti-smoking message during the baseline survey, followed by the threat message one month later in a separate survey. Outcomes will be measured before seeing the anti-smoking message and at 1 month.
  Culturally Tailored Anti-Smoking Messages: Anti-smoking messages will be administered online via a Qualtrics survey.
- Currently Smoking, Three Messages Immediate; Not Currently Smoking, Three Messages Immediate: Participants will receive three anti-smoking messages, followed by the threat message during the baseline survey. Outcomes will be measured before seeing the anti-smoking messages and threat message, immediately after seeing the threat message.
  Culturally Tailored Anti-Smoking Messages: Anti-smoking messages will be administered online via a Qualtrics survey.
- Currently Smoking, Three Messages 1 Week Delay; Not Currently Smoking, Three Messages 1 Week Delay: Participants will receive three anti-smoking messages during the baseline survey, followed by the threat message one week later in a separate survey. Outcomes will be measured before seeing the anti-smoking messages at baseline, immediately after seeing the threat message at 1 week.
  Culturally Tailored Anti-Smoking Messages: Anti-smoking messages will be administered online via a Qualtrics survey.
Period: Overall Study
Arm/Group | Currently Smoking, No Message Condition | Currently Smoking, Single Message Immediate | Currently Smoking, Single Message 1 Week Delay | Currently Smoking, Single Message 1 Month Delay | Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Currently Smoking, Three Messages Immediate | Currently Smoking, Three Messages 1 Week Delay | Currently Smoking, Three Messages 1 Month Delay | Currently Smoking, Three Messages 1 Month Delay Repeat Exposure | Not Currently Smoking, No Message Condition | Not Currently Smoking, Single Message Immediate | Not Currently Smoking, Single Message 1 Week Delay | Not Currently Smoking, Single Message 1 Month Delay | Not Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Not Currently Smoking, Three Messages Immediate | Not Currently Smoking, Three Messages 1 Week Delay | Not Currently Smoking, Three Messages 1 Month Delay | Not Currently Smoking, Three Messages 1 Month Delay Repeat Exposure
Started | 210 | 103 | 113 | 107 | 110 | 107 | 112 | 106 | 107 | 305 | 155 | 146 | 150 | 156 | 146 | 154 | 150 | 154
Completed | 210 | 103 | 75 | 66 | 64 | 107 | 81 | 61 | 65 | 305 | 155 | 109 | 97 | 107 | 146 | 118 | 92 | 101
Not Completed | 0 | 0 | 38 | 41 | 46 | 0 | 31 | 45 | 42 | 0 | 0 | 37 | 53 | 49 | 0 | 36 | 58 | 53
Not completed — Lost to Follow-up | 0 | 0 | 38 | 41 | 46 | 0 | 31 | 45 | 42 | 0 | 0 | 37 | 53 | 49 | 0 | 36 | 58 | 53

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Currently Smoking, No Message Condition | Currently Smoking, Single Message Immediate | Currently Smoking, Single Message 1 Week Delay | Currently Smoking, Single Message 1 Month Delay | Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Currently Smoking, Three Messages Immediate | Currently Smoking, Three Messages 1 Week Delay | Currently Smoking, Three Messages 1 Month Delay | Currently Smoking, Three Messages 1 Month Delay Repeat Exposure | Not Currently Smoking, No Message Condition | Not Currently Smoking, Single Message Immediate | Not Currently Smoking, Single Message 1 Week Delay | Not Currently Smoking, Single Message 1 Month Delay | Not Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Not Currently Smoking, Three Messages Immediate | Not Currently Smoking, Three Messages 1 Week Delay | Not Currently Smoking, Three Messages 1 Month Delay | Not Currently Smoking, Three Messages 1 Month Delay Repeat Exposure | Total
Number analyzed (Participants) | 210 | 103 | 113 | 107 | 110 | 107 | 112 | 106 | 107 | 305 | 155 | 146 | 150 | 156 | 146 | 154 | 150 | 154 | 2591
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.25 (3.35) | 24.37 (3.19) | 24.45 (3.08) | 23.96 (3.20) | 24.32 (3.30) | 24.70 (3.52) | 24.81 (3.26) | 24.41 (3.46) | 24.52 (3.45) | 24.11 (3.22) | 24.75 (3.40) | 24.36 (3.23) | 24.75 (3.53) | 24.29 (3.18) | 23.95 (3.33) | 24.97 (3.20) | 24.27 (3.26) | 24.05 (3.16) | 24.38 (3.29)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 204 | 99 | 110 | 101 | 104 | 104 | 108 | 102 | 98 | 291 | 146 | 136 | 142 | 149 | 138 | 140 | 146 | 149 | 2467
  Male | 6 | 4 | 3 | 6 | 5 | 3 | 3 | 3 | 7 | 14 | 9 | 10 | 7 | 6 | 8 | 14 | 4 | 5 | 117
  Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 18 | 19 | 19 | 20 | 19 | 22 | 18 | 16 | 43 | 21 | 22 | 21 | 20 | 19 | 22 | 21 | 18 | 391
  Not Hispanic or Latino | 177 | 85 | 94 | 88 | 90 | 88 | 90 | 88 | 91 | 262 | 134 | 124 | 129 | 136 | 127 | 132 | 129 | 136 | 2200
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 2 | 4 | 1 | 0 | 2 | 0 | 2 | 1 | 2 | 3 | 2 | 1 | 0 | 0 | 0 | 1 | 24
  Asian | 6 | 4 | 4 | 2 | 3 | 2 | 3 | 1 | 3 | 21 | 10 | 8 | 11 | 11 | 9 | 10 | 10 | 11 | 129
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Black or African American | 38 | 15 | 17 | 13 | 12 | 19 | 19 | 20 | 18 | 20 | 10 | 12 | 13 | 10 | 11 | 14 | 9 | 11 | 281
  White | 141 | 67 | 82 | 79 | 76 | 73 | 70 | 72 | 71 | 219 | 115 | 109 | 111 | 118 | 108 | 109 | 111 | 112 | 1843
  More than one race | 21 | 15 | 7 | 9 | 18 | 13 | 18 | 10 | 13 | 43 | 16 | 13 | 13 | 15 | 17 | 19 | 20 | 17 | 297
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 14
Baseline Intention to Quit Scale [Mean (Standard Deviation); unit: units on a scale] — Sum across 4 items measured on a Likert-scale from 1 to 7.
  Scores range from 4 to 28, higher score indicates higher intention to quit.
  These items were asked among participants who currently smoked. Those who did not smoke currently were not asked these items. Population: These items were asked among participants who currently smoked. Those who did not smoke currently were not asked these items.
  units on a scale
    number analyzed (Participants) | 210 | 103 | 113 | 107 | 110 | 107 | 112 | 106 | 107 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1075
    (all) | 13.78 (8.31) | 13.02 (7.80) | 13.47 (8.65) | 14.33 (8.37) | 13.22 (8.08) | 13.57 (7.20) | 13.91 (7.30) | 13.06 (7.88) | 13.94 (7.77) |  |  |  |  |  |  |  |  |  | 13.61 (7.960)
Intention to Purchase Cigarettes at Baseline [Mean (Standard Deviation); unit: units on a scale] — Single item measure adapted from the Juster Scale measuring intention to purchase cigarettes.
  Scale ranges from 0 (No chance, almost no chance) to 10 (Certain, practically certain), with higher scores indicating greater intentions to purchase cigarettes.
  All participants were asked at baseline.
  units on a scale | 6.76 (3.53) | 7.04 (3.30) | 6.58 (3.68) | 6.51 (3.47) | 6.99 (3.43) | 6.81 (3.30) | 6.96 (3.11) | 7.39 (3.22) | 6.64 (3.58) | 0.29 (0.98) | 0.22 (0.67) | 0.39 (1.13) | 0.28 (0.84) | 0.38 (0.99) | 0.48 (1.47) | 0.33 (1.02) | 0.38 (1.17) | 0.45 (1.25) | 3.04 (3.97)
Susceptibility to smoke cigarettes at baseline [Mean (Standard Deviation); unit: units on a scale] — The susceptibility to smoke cigarettes measure is a sum of responses to 4 items ranging from 0 to 12, higher scores indicating higher susceptibility to smoke.
  Participants who did not smoke currently were asked these questions. Those who currently smoke were not asked these questions. Population: Participants who did not smoke currently were asked these questions. Those who currently smoke were not asked these questions.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 305 | 155 | 146 | 150 | 156 | 146 | 154 | 150 | 154 | 1516
    (all) |  |  |  |  |  |  |  |  |  | 3.19 (2.71) | 2.77 (2.40) | 3.01 (2.84) | 2.93 (2.66) | 3.04 (2.77) | 3.00 (2.90) | 3.11 (2.88) | 2.92 (2.81) | 2.89 (295) | 3.00 (2.76)

OUTCOME MEASURES:

1. Primary Outcome: Intention to Quit Smoking at Follow-up
Description: We used a 4-item scale on intention to quit smoking at baseline and at follow-up (immediate, one-week and one-month) among current smokers only:
  1. I will make an effort to quit smoking in the next 30 days;
  2. I intend to quit smoking in the next 30 days;
  3. I expect to quit smoking in the next 30 days;
  4. How likely is it that you will quit smoking in the next 30 days. Responses ranged on 7-point Likert-like scales. Responses were summed to create a scale for intention to quit (range from 4-28), higher scores indicate higher intention to quit.
Time Frame: Day [0] reported for No-message, single-message immediate, & 3-messages immediate conditions; Week [1] reported for Single-message & 3-messages 1-week delay conditions; Month [1] reported for Single-message & 3-messages 1-month delay conditions
Population: Participants who were currently not smoking were not asked intentions to quit questions
  Participants in the no-message and immediate conditions were not asked post-test intentions to quit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Currently Smoking, No Message Condition | Currently Smoking, Single Message Immediate | Currently Smoking, Single Message 1 Week Delay | Currently Smoking, Single Message 1 Month Delay | Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Currently Smoking, Three Messages Immediate | Currently Smoking, Three Messages 1 Week Delay | Currently Smoking, Three Messages 1 Month Delay | Currently Smoking, Three Messages 1 Month Delay Repeat Exposure | Not Currently Smoking, No Message Condition | Not Currently Smoking, Single Message Immediate | Not Currently Smoking, Single Message 1 Week Delay | Not Currently Smoking, Single Message 1 Month Delay | Not Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Not Currently Smoking, Three Messages Immediate | Not Currently Smoking, Three Messages 1 Week Delay | Not Currently Smoking, Three Messages 1 Month Delay | Not Currently Smoking, Three Messages 1 Month Delay Repeat Exposure
Number analyzed (Participants) | 0 | 0 | 75 | 66 | 63 | 0 | 80 | 60 | 65 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
units on a scale |  |  | 11.8 (8.5) | 11.0 (9.0) | 14.4 (8.1) |  | 9.9 (7.8) | 11.1 (8.4) | 14.4 (7.9) |  |  |  |  |  |  |  |  |

2. Primary Outcome: Intention to Purchase Cigarettes
Description: The Juster scale was used to measure intention to purchase cigarettes at baseline and at one-month follow-up.
  Participants were asked, "How likely are you to purchase cigarettes in the next 6 months?" Responses ranged from 0=No chance, almost no chance (1 in 100) to 10=Certain, practically certain (99 in 100).
  Higher values reflect higher intention to purchase.
Time Frame: as for outcome 1
Population: Participants in the no-message condition and immediate conditions were not asked post-test intention to purchase.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Currently Smoking, No Message Condition | Currently Smoking, Single Message Immediate | Currently Smoking, Single Message 1 Week Delay | Currently Smoking, Single Message 1 Month Delay | Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Currently Smoking, Three Messages Immediate | Currently Smoking, Three Messages 1 Week Delay | Currently Smoking, Three Messages 1 Month Delay | Currently Smoking, Three Messages 1 Month Delay Repeat Exposure | Not Currently Smoking, No Message Condition | Not Currently Smoking, Single Message Immediate | Not Currently Smoking, Single Message 1 Week Delay | Not Currently Smoking, Single Message 1 Month Delay | Not Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Not Currently Smoking, Three Messages Immediate | Not Currently Smoking, Three Messages 1 Week Delay | Not Currently Smoking, Three Messages 1 Month Delay | Not Currently Smoking, Three Messages 1 Month Delay Repeat Exposure
Number analyzed (Participants) | 0 | 0 | 75 | 66 | 64 | 0 | 81 | 61 | 65 | 0 | 0 | 109 | 97 | 107 | 0 | 114 | 92 | 101
units on a scale |  |  | 5.5 (3.8) | 5.7 (3.7) | 4.2 (3.8) |  | 5.9 (3.3) | 5.7 (3.5) | 3.9 (3.4) |  |  | 0.4 (1.4) | 0.2 (0.5) | 0.4 (1.2) |  | 0.2 (0.5) | 0.3 (1.1) | 0.4 (1.3)

3. Primary Outcome: Susceptibility to Smoke Cigarettes
Description: Susceptibility to smoke cigarettes were measured using four-items:
  1. Have you ever been curious about smoking a cigarette?
  2. Do you think you will smoke a cigarette in the next year?
  3. Do you think that you will try a cigarette soon?
  4. If one of your best friends were to offer you a cigarette, would you smoke it? Responses ranged on 4-point Likert-like scales.
  Responses were summed to create a scale for susceptibility to smoke cigarettes (range from 0-12). This was only measured among participants who did not currently smoke.
  Higher scores indicate increased susceptibility to smoke cigarettes.
Time Frame: as for outcome 1
Population: This was only measured among participants who did not currently smoke.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Currently Smoking, No Message Condition | Currently Smoking, Single Message Immediate | Currently Smoking, Single Message 1 Week Delay | Currently Smoking, Single Message 1 Month Delay | Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Currently Smoking, Three Messages Immediate | Currently Smoking, Three Messages 1 Week Delay | Currently Smoking, Three Messages 1 Month Delay | Currently Smoking, Three Messages 1 Month Delay Repeat Exposure | Not Currently Smoking, No Message Condition | Not Currently Smoking, Single Message Immediate | Not Currently Smoking, Single Message 1 Week Delay | Not Currently Smoking, Single Message 1 Month Delay | Not Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Not Currently Smoking, Three Messages Immediate | Not Currently Smoking, Three Messages 1 Week Delay | Not Currently Smoking, Three Messages 1 Month Delay | Not Currently Smoking, Three Messages 1 Month Delay Repeat Exposure
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 305 | 155 | 108 | 97 | 107 | 146 | 114 | 92 | 101
units on a scale |  |  |  |  |  |  |  |  |  | 3.0 (2.6) | 2.7 (2.4) | 2.2 (2.7) | 2.8 (2.5) | 2.5 (2.7) | 3.0 (2.9) | 1.9 (2.8) | 2.6 (2.6) | 2.8 (3.0)

4. Secondary Outcome: Receptivity to Marketing
Description: Receptivity to marketing was measured using 2 items:
  1. Tobacco companies should have the same rights to advertise as other companies.
  2. Are you open to using or wearing something with a tobacco company logo or picture on it? Response options range from 1 (strongly agree) to 5 (strongly disagree)
  The scale is a sum of the responses to these items, the scale ranges from 2 to 10, with lower scores indicating greater receptivity to marketing.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Currently Smoking, No Message Condition | Currently Smoking, Single Message Immediate | Currently Smoking, Single Message 1 Week Delay | Currently Smoking, Single Message 1 Month Delay | Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Currently Smoking, Three Messages Immediate | Currently Smoking, Three Messages 1 Week Delay | Currently Smoking, Three Messages 1 Month Delay | Currently Smoking, Three Messages 1 Month Delay Repeat Exposure | Not Currently Smoking, No Message Condition | Not Currently Smoking, Single Message Immediate | Not Currently Smoking, Single Message 1 Week Delay | Not Currently Smoking, Single Message 1 Month Delay | Not Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Not Currently Smoking, Three Messages Immediate | Not Currently Smoking, Three Messages 1 Week Delay | Not Currently Smoking, Three Messages 1 Month Delay | Not Currently Smoking, Three Messages 1 Month Delay Repeat Exposure
Number analyzed (Participants) | 210 | 103 | 75 | 66 | 64 | 107 | 81 | 61 | 65 | 304 | 155 | 109 | 97 | 107 | 146 | 114 | 92 | 101
units on a scale | 6.3 (2.5) | 6.1 (2.6) | 6.4 (2.5) | 6.6 (2.5) | 6.8 (2.4) | 6.5 (2.5) | 6.7 (2.6) | 6.3 (2.6) | 7.2 (2.5) | 8.3 (1.7) | 8.5 (1.5) | 8.4 (1.5) | 8.4 (1.6) | 8.4 (1.4) | 8.6 (1.4) | 8.3 (1.6) | 8.2 (1.7) | 8.4 (1.4)

5. Secondary Outcome: Tobacco Industry Attitudes
Description: Tobacco industry attitudes were measured using 3 items:
  1. I would like to see cigarette companies go out of business.
  2. I would not work for a cigarette company.
  3. How much do you like cigarette companies.
  Response options for items 1 and 2 were from 1 (Strongly agree) to 5 (Strongly disagree). Response options for item 3 were from 1 (Dislike strongly) to 5 (Like strongly). Response options were summed across these 3 items to create the tobacco industry attitudes scale.
  Values range from 3 to 15, with lower scores indicating stronger anti-industry sentiment.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Currently Smoking, No Message Condition | Currently Smoking, Single Message Immediate | Currently Smoking, Single Message 1 Week Delay | Currently Smoking, Single Message 1 Month Delay | Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Currently Smoking, Three Messages Immediate | Currently Smoking, Three Messages 1 Week Delay | Currently Smoking, Three Messages 1 Month Delay | Currently Smoking, Three Messages 1 Month Delay Repeat Exposure | Not Currently Smoking, No Message Condition | Not Currently Smoking, Single Message Immediate | Not Currently Smoking, Single Message 1 Week Delay | Not Currently Smoking, Single Message 1 Month Delay | Not Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Not Currently Smoking, Three Messages Immediate | Not Currently Smoking, Three Messages 1 Week Delay | Not Currently Smoking, Three Messages 1 Month Delay | Not Currently Smoking, Three Messages 1 Month Delay Repeat Exposure
Number analyzed (Participants) | 209 | 103 | 75 | 66 | 64 | 107 | 81 | 61 | 64 | 304 | 154 | 109 | 97 | 107 | 146 | 114 | 92 | 101
units on a scale | 8.1 (3.4) | 8.2 (3.4) | 7.8 (3.4) | 7.6 (3.5) | 7.1 (2.8) | 7.4 (3.5) | 8.0 (3.3) | 7.8 (3.3) | 6.7 (3.2) | 5.0 (2.2) | 4.8 (1.8) | 4.5 (1.8) | 4.7 (1.8) | 4.6 (2.0) | 4.8 (2.1) | 4.9 (2.2) | 4.8 (2.1) | 4.6 (2.0)

6. Secondary Outcome: Tobacco Industry Beliefs
Description: Industry beliefs were measured using 4 items:
  Cigarette companies lie. Cigarette companies target teens to replace smokers who die. Cigarette companies deny that cigarettes cause cancer and other harmful diseases.
  Cigarette companies deny that cigarettes are addictive.
  Response options were from 1 (Strongly agree) to 5 (Strongly disagree).
  Responses were summed across these 4 items to create the tobacco industry beliefs scale. Values ranges from 4 to 20, with lower scores indicating stronger anti-industry sentiment.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Currently Smoking, No Message Condition | Currently Smoking, Single Message Immediate | Currently Smoking, Single Message 1 Week Delay | Currently Smoking, Single Message 1 Month Delay | Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Currently Smoking, Three Messages Immediate | Currently Smoking, Three Messages 1 Week Delay | Currently Smoking, Three Messages 1 Month Delay | Currently Smoking, Three Messages 1 Month Delay Repeat Exposure | Not Currently Smoking, No Message Condition | Not Currently Smoking, Single Message Immediate | Not Currently Smoking, Single Message 1 Week Delay | Not Currently Smoking, Single Message 1 Month Delay | Not Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Not Currently Smoking, Three Messages Immediate | Not Currently Smoking, Three Messages 1 Week Delay | Not Currently Smoking, Three Messages 1 Month Delay | Not Currently Smoking, Three Messages 1 Month Delay Repeat Exposure
Number analyzed (Participants) | 210 | 102 | 75 | 66 | 64 | 106 | 81 | 61 | 63 | 304 | 153 | 109 | 97 | 107 | 145 | 113 | 92 | 101
units on a scale | 11.7 (4.5) | 11.7 (4.9) | 10.9 (4.4) | 11.1 (4.7) | 10.4 (4.3) | 11.0 (4.2) | 11.4 (4.0) | 10.5 (4.5) | 10.5 (4.4) | 8.9 (3.7) | 8.3 (3.5) | 8.9 (3.5) | 8.9 (3.2) | 8.7 (3.4) | 8.5 (3.4) | 8.9 (3.3) | 9.2 (3.6) | 8.8 (3.3)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Currently Smoking, No Message Condition | Currently Smoking, Single Message Immediate | Currently Smoking, Single Message 1 Week Delay | Currently Smoking, Single Message 1 Month Delay | Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Currently Smoking, Three Messages Immediate | Currently Smoking, Three Messages 1 Week Delay | Currently Smoking, Three Messages 1 Month Delay | Currently Smoking, Three Messages 1 Month Delay Repeat Exposure | Not Currently Smoking, No Message Condition | Not Currently Smoking, Single Message Immediate | Not Currently Smoking, Single Message 1 Week Delay | Not Currently Smoking, Single Message 1 Month Delay | Not Currently Smoking, Single Message 1 Month Delay, Repeated Exposure | Not Currently Smoking, Three Messages Immediate | Not Currently Smoking, Three Messages 1 Week Delay | Not Currently Smoking, Three Messages 1 Month Delay | Not Currently Smoking, Three Messages 1 Month Delay Repeat Exposure
All-Cause Mortality (participants affected / at risk) | 0/210 | 0/103 | 0/113 | 0/107 | 0/110 | 0/107 | 0/112 | 0/106 | 0/107 | 0/305 | 0/155 | 0/146 | 0/150 | 0/156 | 0/146 | 0/154 | 0/150 | 0/154
Serious Adverse Events (participants affected / at risk) | 0/210 | 0/103 | 0/113 | 0/107 | 0/110 | 0/107 | 0/112 | 0/106 | 0/107 | 0/305 | 0/155 | 0/146 | 0/150 | 0/156 | 0/146 | 0/154 | 0/150 | 0/154
Other Adverse Events (participants affected / at risk) | 0/210 | 0/103 | 0/113 | 0/107 | 0/110 | 0/107 | 0/112 | 0/106 | 0/107 | 0/305 | 0/155 | 0/146 | 0/150 | 0/156 | 0/146 | 0/154 | 0/150 | 0/154

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT05499520/Prot_SAP_000.pdf